CLINICAL TRIAL: NCT06596915
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Preliminary Efficacy of BA1302 in Patients With Advanced Solid Malignancies
Brief Title: Safety and Efficacy of BA1302 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA1302/CT-CHN-101
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer; Pancreatic Adenocarcinoma; Breast Cancer; Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BA1302 (Experimental)
  Interventions: Drug: BA1302

INTERVENTIONS:
Drug: BA1302 — BA1302 administered intravenously

SUMMARY:
This is a first-in-human (FIH), multicenter, open-label Phase I study to evaluate the safety, tolerability, PK profile, immunogenicity, and preliminary efficacy of BA1302 in patients with advanced solid malignancies. The study includes a dose-escalation phase (Part A) and a dose-expansion phase (Part B).

ELIGIBILITY:
Inclusion Criteria:

* 1. Metastatic or unresectable solid malignancy that is histologically or cytologically confirmed. Patients who have progressed on or after standard therapy, or are intolerant of standard therapy, or have no appropriate standard therapy available.

  1. Part A: Advanced malignant solid tumors;
  2. Part B: Metastatic melanoma, Advanced breast cancer, Advanced Non-small cell lung cancer (NSCLC), Advanced pancreatic adenocarcinoma.
* 2.Participants should be able to provide adequate tumor tissue for biomarker analysis
* 3.ECOG Performance Status ≤ 1.
* 4.Measurable disease per Response Evaluation Criteria for Solid Tumors version 1.1 (RECIST v1.1)

Exclusion Criteria:

* 1. Malignant disease within 5 years prior to the first dose of investigational drug other than that being treated in this study. Except completely resected basal cell carcinoma, cutaneous squamous cell skin carcinoma and papillary thyroid carcinoma and completely resected carcinoma in situ of any type.
* 2. Received any chemotherapy, radiotherapy, targeted therapy, cell therapy, immunotherapy, ADC medication or other anti-cancer treatment within 28 days prior to the first dose.
* 3.History of severe hypersensitivity reactions to any ingredient of study drugs.
* 4.Pregnant or lactating women.
* 5.Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | Up to 21 days
adverse events | Through 28 days after the last study treatment

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) from time zero to the last quantifiable concentration (AUC0-t) | Up to approximately 1 years
AUC from time zero to infinity (AUC0-inf) | Up to approximately 1 years
Maximum serum concentration (Cmax) | Up to approximately 1 years
Elimination half-life (t1/2) | Up to approximately 1 years
Area under the concentration-time curve (AUC) at steady state | Up to approximately 1 years
Incidence of anti-drug antibodies (ADA) | Up to approximately 1 years
Objective response rate (ORR) | Up to approximately 1 years
Duration of objective response (DOR) | Up to approximately 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China